CLINICAL TRIAL: NCT07137637
Title: Phase 1 Dose Escalation and Expansion Study of HPB-092 to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy in Patients With Relapsed or Refractory Acute Myeloid Leukemia (RR-AML)
Brief Title: HPB-092 for the Treatment of Relapsed and Refractory Acute Myeloid Leukemia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Polymed Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HPB-092-CN101
Record Dates: First submitted 2025-07-31; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Relapsed and Refractory Acute Myeloid Leukemia (RR-AML)
Keywords: Interleukin-1 receptor-associated kinase 4 (IRAK4); SF3B1; U2AF1; FLT3 mutation; FLT3 inhibitor; IRAK4 inhibitor; Dual Kinase Inhibitor FLT3 and IRAK4; Relapsed and Refractory Acute Myeloid Leukemia (RR-AML); Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Intervention Model Description: This Phase 1 study includes two parts: Part A for dose escalation and Part B for dose expansion, involving single or multiple doses.
  In Part A, up to 5 dose levels will be evaluated in RR-AML patients with FLT3 mutations. The starting dose is 30 milligrams (mg) administered twice daily (BID).
  In Part B, once the recommended expansion doses (RED) are established based on the maximum tolerated dose (MTD) from Part A, RR-AML patients with FLT3 mutations and/or spliceosome mutations in SF3B1 or U2AF1 will be enrolled across up to 3 dose levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HPB-092 Monotherapy - Dose Escalation and Expansion (Experimental): RR-AML patients receive HPB-092 tablet monotherapy BID daily. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: HPB-092 tablet

INTERVENTIONS:
Drug: HPB-092 tablet — HPB-092 is formulated as a tablet for oral administration, taken twice daily (BID) over consecutive 28-day cycles. This novel small molecule selectively inhibits both FLT3 and interleukin-1 receptor-associated kinase 4 (IRAK4). IRAK4 plays a crucial role in the toll-like receptor (TLR) and interleukin-1 receptor (IL-1R) signaling pathways, which are frequently dysregulated in acute myeloid leukemia (AML) and other malignancies.

SUMMARY:
HPB-092 effectively inhibits Fms-like tyrosine kinase 3 (FLT3) mutants with comparable or superior potency to approved FLT3 inhibitors and demonstrates improved selectivity, potentially reducing toxicity. Its highly selective and potent inhibition of Interleukin-1 Receptor-Associated Kinase 4 (IRAK4) may provide additional therapeutic benefits that could enhance treatment efficacy and durability for patients with relapsed or refractory acute myeloid leukemia (RR-AML), further improving clinical outcomes in this population. HPB-092 also has a favorable safety profile, with no major risks identified in preclinical studies.

Phas 1 Study Outline:

1. This is a multicenter, open-label, phase 1 study to evaluate the safety and efficacy of oral HPB-092 as monotherapy in patients with RR-AML.
2. The study aims to assess safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy.
3. It consists of two parts: Part A for dose escalation and Part B for dose expansion, involving single or multiple doses.
4. Patients must be diagnosed with morphologically documented RR-AML according to World Health Organization (WHO) 2022 criteria.
5. Baseline assessments will include RR-AML with FLT3 mutations, spliceosome mutations in SF3B1 and U2AF1, as well as other biomarkers, which will be monitored throughout the study.

DETAILED DESCRIPTION:
HPB-092 - A Novel Dual Selective Kinase Inhibitor of FLT3 and IRAK4:

Multiple FLT3 inhibitors have been approved for clinical use in acute myeloid leukemia (AML). However, many patients do not benefit from these therapies due to toxicities and resistance. IRAK4 is a serine/threonine kinase involved in innate immune signaling. Overexpression of IRAK4-particularly the long isoform (IRAK4-L)-is common in most AML cases and is associated with poor prognosis and resistance to FLT3 inhibitors, suggesting that dual inhibition of FLT3 and IRAK4 may provide therapeutic benefits.

HPB-092 is an effective dual inhibitor of FLT3 and IRAK4, exhibiting high selectivity, favorable absorption, distribution, metabolism, and excretion (ADME) properties, as well as strong anti-leukemic efficacy. It also has a broader safety window in non-clinical studies compared to existing FLT3 inhibitors. Given its potential to address unmet medical needs in RR-AML patients, particularly those resistant to existing FLT3 inhibitors, HPB-092 warrants further clinical investigation.

Primary Objective and Endpoints:

The primary objective of this Phase 1 study is to evaluate the safety and tolerability of HPB-092 monotherapy in patients with RR-AML. The primary endpoints will include assessments of adverse events (AEs), treatment-emergent adverse events (TEAEs), dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD).

Secondary Objectives:

The secondary objectives of this Phase 1 study are as follows:

1. To characterize the pharmacokinetic profile of HPB-092.
2. To determine the minimum safe dose and Biologically Effective Dose (BED) of HPB-092.
3. To evaluate the anti-leukemic activity of various dose levels of HPB-092.
4. To establish the Recommended Phase 2 Dose (RP2D) of HPB-092 in patients with RR-AML.

Exploratory Objectives:

The exploratory objectives will focus on the clinical pharmacology of HPB-092, including the identification of potential biomarkers to predict the response to HPB-092 in AML patients.

Part A Dosing Protocol:

HPB-092 is available in tablet form, with two strengths: 10 and 40 milligrams (mg). In Part A of the dose escalation, the starting dose will be 30 mg administered twice daily (BID), with subsequent dose escalations planned up to five dose levels. This approach aims to determine the Recommended Expansion Dose (RED) for the Part B dose expansion cohorts. Each treatment cycle will last 28 days and may be repeated in the absence of DLT or other toxicities, as determined by the investigator. Patients who derive clinical benefit from the study treatment may continue for up to two years from the initiation of the study drug or until one or more treatment discontinuation criteria are met.

In each dose escalation cohort, patients with RR-AML will be enrolled at the designated dose. Dose escalation will follow modified 3+3 rules, with DLT assessed during the first cycle. Escalation to the next dose level will occur as soon as the safety of the current dose is confirmed in a Cohort Review Meeting. The dose and schedule of HPB-092 administered to each patient will be documented on the appropriate form for each cycle.

Part B Dosing Protocol:

The Part B expansion, consisting of up to 3 dose levels, will begin once the recommended expansion doses (RED) is established based on the maximum tolerated dose (MTD) determined in Part A. This Part B expansion aims to further evaluate the efficacy, safety, pharmacokinetics (PK), and pharmacodynamics (PD) of HPB-092, as well as to determine the recommended phase II dose (RP2D). The RP2D will be reviewed by a Cohort Review Meeting based on the results from Part B, considering all aspects of safety, tolerability, biological activity, pharmacokinetics, and preliminary efficacy in the trial population. The intent of the RP2D is to establish recommended dose levels and dosing intervals for the Phase II study, maximizing the potential for clinical benefit while minimizing the risk of toxicity. The Cohort Review Meeting may request the recruitment of additional patients at any previously explored or intermediate dose level to make an appropriate RP2D decision for the Phase 2 study.

Ethical Conduct of the Study:

The study will be conducted in accordance with the protocol, ICH guidelines, and applicable regulations governing clinical study conduct. Additionally, it will adhere to ethical principles derived from the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrollment in the study:

1. The patient must have a diagnosis of morphologically documented relapsed or refractory acute myeloid leukemia (AML) according to the World Health Organization (WHO) 2022 criteria, and must meet one of the following conditions:

   Relapsed Disease: Bone marrow blasts ≥ 5%; or Reappearance of blasts in the peripheral blood in at least two separate samples taken at least one week apart; or Development of extramedullary disease. Refractory Disease: Failure to achieve CR, CRh, or CRi at the response landmark (e.g., after 2 courses of intensive induction therapy), or Failure to achieve remission by a defined landmark, e.g., 180 days after initiation of less intensive therapy.
2. The patients should have a stable transfusion requirement prior to enrollment as specified in the protocol.
3. Male or non-pregnant, non-lactating female patients aged 18 years or older.
4. The patient is not suitable for other known therapies that have clinical benefits for the disease.
5. Life expectancy of ≥12 weeks, and Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
6. Renal Function: Serum creatinine <1.5× the upper limit of normal (ULN) or Estimated creatinine clearance ≥ 60 mL/min as calculated using a standard method [Cockcroft-Gault formula, Modification of Diet in Renal Disease (MDRD) equation, or estimated glomerular filtration rate (eGFR) calculation]. Liver Function: Total serum bilirubin ≤1.5× ULN unless the patient has liver involvement by the primary disease (≤3× ULN); and AST and ALT ≤2.5× ULN unless the patient has hepatic metastasis (≤5× ULN). Cardiac Function: Left ventricular ejection fraction (LVEF) >50% as measured by echocardiogram or MUGA scan.
7. Acute effects of any prior therapy must be resolved to baseline severity or Grade ≤ 1 per CTCAE v5.0, except for adverse events (AEs) that do not constitute a safety risk according to the investigator's judgment.
8. For females of childbearing potential, a serum pregnancy test must be negative within 7 days before enrollment.
9. Male and female patients of childbearing potential who are at risk for pregnancy must agree to use at least two highly effective methods of contraception throughout the study and for at least 90 days (or 180 days if required by local regulations) after the last dose of the assigned treatment.
10. The interval from prior treatment to the time of study drug administration must be at least 2 weeks for cytotoxic agents (except hydroxyurea given for controlling blast cells), or at least 5 half-lives for prior experimental agents or noncytotoxic agents.
11. The patient must have the ability to understand and be willing to sign the informed.

Exclusion Criteria:

Patients with any of the following characteristics/conditions will not be able to enroll in the study:

1. Diagnosed with acute promyelocytic leukemia (APL) or BCR-ABL-positive leukemia.
2. The patient has had a malignancy other than AML within the past five years as specified in the protocol.
3. The patient has persistent non-hematological toxicities of ≥ Grade 2 (per CTCAE v5.0) from prior treatment.
4. History of Hematopoietic Stem Cell Transplant (HSCT) as specified in the protocol.
5. The patient has clinically active central nervous system (CNS) leukemia.
6. The patient has a disseminated intravascular coagulation (DIC) abnormality.
7. Recent surgery or radiation therapy as specified in the protocol.
8. History of Class 3 or more severe heart failure according to NYHA classification, or left ventricular ejection fraction (LVEF) below 45%, or Fridericia-corrected QT interval (QTcF) > 450 ms at screening.
9. The patient has hypokalemia or hypomagnesemia at screening.
10. The patient requires treatment with drugs that are strong inhibitors or inducers of CYP3A4 or P-glycoprotein (P-gp) as specified in the protocol.
11. Active graft-versus-host disease (GVHD) and immunosuppressive treatment as specified in the protocol.
12. Use of systemic corticosteroids or immunosuppressive drugs as specified in the protocol.
13. The patient is known to be infected with human immunodeficiency virus (HIV), active hepatitis B or C, or other active hepatic disorders. The patient has an active uncontrolled infection.
14. The patient has any condition that, in the investigator's opinion, makes the patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-09-14 (Estimated); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
Adverse Events and Treatment-Emergent Adverse Events [Safety and Tolerability] | From the first dose (Cycle 1 day 1) of HPB-092 treatment until 28 days after the completion of treatment, or after early termination or withdrawal from the study, with a duration of up to 24 months
  Adverse events (AEs) and treatment-emergent adverse events (TEAEs) will be measured by the number of participants who have received at least one dose of HPB-092. All AEs and TEAEs will be assessed and reported in accordance with the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Dose-Limiting Toxicity [Safety and Tolerability] | Days 1-28 of the first cycle (each cycle is 28 days)
  The Dose-Limiting Toxicity (DLT) will be determined based on the first cycle (Days 1-28) of HPB-092 in RR-AML patients. Reviews of DLT for dose escalation decisions will be conducted for each completed dose level. Dose escalation decisions will require full safety data review of all subjects who completed Cycle 1 (Days 1-28) or discontinued due to a suspected DLT within Cycle 1 (Days 1-28).
Maximum Tolerated Dose [Safety and Tolerability] | Days 1-28 of the first cycle (each cycle is 28 days)
  The Maximum Tolerated Dose (MTD) is defined as the highest dose level at which ≤1 of 6 evaluable RR-AML subjects (≤33%) experience a DLT during Cycle 1 (Days 1-28). If ≥2 DLTs occur at a given dose level, the preceding dose will be expanded to 6 additional subjects for MTD confirmation. All subjects must complete the DLT observation period (Cycle 1, Days 1-28) to be evaluable; early discontinuations due to non-DLT reasons will be replaced.

SECONDARY OUTCOMES:
Characterization of the pharmacokinetic (PK) parameters of HPB-092, measured by the maximum plasma concentration (Cmax), in AML patients. | Up to 24 months
  Maximum plasma concentration (Cmax) in AML patients
Characterization of the pharmacokinetic (PK) parameters of HPB-092, measured by Time to maximum plasma concentration (Tmax), in AML patients | Up to 24 months
  Time to maximum plasma concentration (Tmax) in AML patients
Characterization of the pharmacokinetic (PK) parameters of HPB-092, measured by Area under the plasma concentration versus time curve (AUC) [0-24], in AML patients | Up to 24 months
  Area under the plasma concentration-time curve from 0 to 24 hours in AML patients
Characterization of the pharmacokinetic (PK) parameters of HPB-092, measured by Area under the plasma concentration versus time curve (AUC) [0-inf], in AML patients | Up to 24 months
  Area under the plasma concentration-time curve from 0 to infinity in AML patients
Characterization of the pharmacokinetic (PK) parameters of HPB-092, measured by Plasma terminal elimination half-life (T1/2), in AML patients | Up to 24 months
  Plasma terminal elimination half-life (T1/2) in AML patients
Characterization of the pharmacokinetic (PK) parameters of HPB-092, measured by the plasma clearance (CL), in AML patients. | Up to 24 months
  Calculation of the clearance (CL) of HPB-092 in AML patients, determined by the plasma drug concentration-time curve area under the curve (AUC) and the administered dose.
Assessment of the Efficacy of Clinical Response to HPB-092 Monotherapy in AML Patients. | up to 24 months
  Definitions for treatment response will follow the 2022 recommendations for the diagnosis and management of AML in adults from an international expert panel on behalf of the European LeukemiaNet (ELN).
  The clinical response to HPB-092 monotherapy in AML patients will be evaluated by determining the percentage of patients who achieve any of the following outcomes: complete remission (CR), complete remission with partial hematologic recovery (CRh), complete remission with incomplete hematologic recovery (CRi). The Disease Control Rate (DCR) is defined as the confirmed remission rate, encompassing all complete responses (CR + CRh + CRi) in AML patients.
Assessment of the Duration of Response to HPB-092 Monotherapy in AML Patients. | Up to 24 months
  Assessed by the Duration of Response (DoR) to HPB-092 monotherapy in AML patients. The DoR is defined as the time from the first documentation of a complete response (CR, CRh, or CRi) until the first occurrence of disease progression or relapse in AML patients.
Assessment of the Time to Response to HPB-092 Monotherapy in AML Patients. | Up to 24 months
  Time to Response (TTR) is defined as the duration from the initiation of HPB-092 monotherapy to the first documentation of a clinical response (including CR, CRh, or CRi) in AML patients.
Determination of the Recommended Phase 2 Dose (RP2D) of HPB-092 Monotherapy in AML Patients. | Up to 24 months
  The Recommended Phase 2 Dose (RP2D) will be determined during the Cohort Review Meeting, taking into account all aspects of safety, tolerability, biological activity, pharmacokinetics, and preliminary efficacy within the trial population. The aim of establishing an RP2D is to identify a dose and schedule that optimize the potential for clinical benefit while minimizing the risk of toxicity in AML Patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, MD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, China

IPD SHARING:
Plan to Share IPD: No